CLINICAL TRIAL: NCT04609085
Title: SARS-COV2 Pandemic Serosurvey in a Rare Disease Population
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000210; 000210-I
Record Dates: First submitted 2020-10-29; First posted 2020-10-30 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: SARS-COV2 Virus
Keywords: COVID-19; Rare Diseases; Antibodies; Natural History
MeSH Terms: conditions — COVID-19; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Rare Diseases: Participants with history of rare disease

SUMMARY:
Background:

The SARS-COV2 outbreak has had a major impact on the economy and society. Researchers want to learn how widespread the infection is in the rare disease community. To do this, they will get blood samples from people with rare diseases. They will use at-home sampling. This will allow them to get samples from people across a wide area.

Objective:

To estimate the proportion of people with rare diseases who have SARS-COV2 antibodies in the National Center for the Advancement of Translational Sciences Rare Disease Clinical Research Network (RDCRN) Rare Diseases Survey over time.

Eligibility:

People under age 90 who have a rare disease and have taken part in the Cincinnati Children s Hospital Medical Center (CCHMC) protocol# 2020-0299.

Design:

RDCRN will tell CCHMC participants about this NIH study. RDCRN will only reach out to those who agreed to be contacted for future studies. They will be contacted by phone and email.

Participants will have a virtual visit to collect data. It will take place over the phone.

Participants will be sent a home kit to collect a blood sample. The kit contains gauze, a lancet, bandages, a collection device, and instructions. They will also be given shipping materials. They will give up to 80ul of blood. They will ship the sample back to NIH.

Participants will complete a survey. It can be done online or over the phone.

Participation will last for 1 week....

DETAILED DESCRIPTION:
It has been demonstrated that respiratory virus outbreaks and pandemics, such as influenza, SARS, MERS, and now the newly emerged SARS-COV2 virus, have a major impact on morbidity and mortality worldwide, as well as having devastating global economic and societal impact. During these outbreaks it is critical to gain a rapid understanding of the exposures and immunity in the general population. Current ongoing serosurvey efforts to estimate the prevalence of infection/exposure are focused on the general population, but these estimates may not be applicable to individuals living with rare diseases. An effort to identify the impact of this pandemic on this community is underway in the Rare Disease Clinical Research Network (RDCRN) led by the Data Management and Coordinating Center (DMCC) at Cincinnati Children s Hospital Medical Center (CCHMC) supported by NCATS. Through a survey they are attempting to evaluate infection rates and impact on those with rare diseases. In this study we propose to enroll a subset of the individuals participating in the RDCRN study to collect blood for SARS-Cov-2 antibody testing. This will allow us to add a biological marker to confirm infection/exposure and further our understanding of how widespread this infection is in the rare diseae community.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. <90 years of age.
  2. Participant in CCHMC Protocol# 2020-0299.
  3. Will have expressed interest in discussing this study with us when contacted by CCHMC Protocol# 2020-0299 study team.
  4. Willing and able to complete a verbal telephone consent or, has a parent/guardian or Legally Authorized Representative (LAR) able to complete the consent.
  5. Willing to undergo home blood sampling procedures.
  6. Willing to have blood samples stored for future research.

EXCLUSION CRITERIA:

1. Unable to provide consent and/or does not have a parent, guardian, or LAR to provide consent
2. Any condition or event that, in the PI s opinion, may substantially increase the risk associated with study participation or compromise the study s scientific objectives. Conditions that exclude a subject are considered to be unlikely, but an example would include having an acute respiratory infection that would make it unsafe to obtain blood samples.
3. Not willing to have blood samples stored for future research.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are enrolled in CCHMC protocol# 2020-0299 Impact of COVID-19 on People Living with Rare Diseases and their Families.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
To estimate the proportion of people with rare diseases who have detectable antibodies to SARS-COV2 in the NCATS RDCRN Rare Diseases Survey. | 2 years
  Anti-SARS-COV2 IgG, IgA, and IgM measured by ELISA

SECONDARY OUTCOMES:
To estimate the proportion of detectable antibodies across specific categories of rare diseases (e.g., people who live with rare diseases characterized by immune compromise vs. people with hyper-reactivity of the immune system). | 2 years
  Variation in the Observed-to-expected ratio of people with detectable Anti-SARS-COV2 IgG, IgA, and IgM measured by ELISA (seroprevalent cases), across subgroups of people with different categories of rare diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
.IDP will be made available through the NCI Seronet and clinical trials.gov. IDP that underlies the results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be shared starting a maximum of 1 year after publication.
Access Criteria: The IPD will be available publicly.